CLINICAL TRIAL: NCT02826018
Title: A Phase 1/2, Randomized, Single-Blind, Placebo-Controlled, Single-Ascending and Multiple-Ascending Dose, Safety, Tolerability, Pharmacokinetics, and Antiviral Efficacy Study of Subcutaneously Administered ALN-HBV in Healthy Adult Subjects and Non-cirrhotic Patients With Chronic Hepatitis B Virus (HBV) Infection
Brief Title: A Study of ALN-HBV in Healthy Adult Volunteers and Non-cirrhotic Patients With Chronic Hepatitis B Virus (HBV) Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALN-HBV-001
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis B; Chronic Hepatitis B; Hepatitis B, Chronic; Hepatitis B Infection; HBV
Keywords: RNAi therapeutic; Hepatitis B; Chronic Hepatitis B; Hepatitis B, Chronic; Hepatitis B Infection; HBV
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALN-HBV (Active Comparator)
  Interventions: Drug: ALN-HBV
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: ALN-HBV — Ascending doses of ALN-HBV by subcutaneous (sc) injection
  Arms: ALN-HBV
Drug: Sterile Normal Saline (0.9% NaCl) — Calculated volume to match active comparator
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics of ALN-HBV in healthy adult volunteers and patients with chronic hepatitis B virus (HBV) infection. In addition, the study will assess antiviral efficacy of ALN-HBV in patients with HBV.

DETAILED DESCRIPTION:
The study has 3 parts. Part A is a single ascending dose (SAD) study in healthy volunteers. Part B is a single ascending dose study (SAD) in patients with HBV infection. Part C is a multiple ascending dose study (MAD) in patients with HBV infection.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* 18 to 65 years inclusive
* Women of child-bearing potential must have a negative pregnancy test, cannot be breast feeding, and must be willing to use a highly effective method of contraception
* Agrees not to donate blood during the duration of the study
* Willing to comply with the study requirements and to provide written informed consent

Additional inclusion criteria for patients with HBV infection:

* Body mass index (BMI) ≥18.0 kg/m2
* Must be on a stable regimen of entecavir or tenofovir

Exclusion Criteria:

All subjects:

* Any uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with participation in the clinical study, and/or put the subject at significant risk
* Subjects with a history of serious mental illness
* Active infection with human immunodeficiency virus (HIV) infection, hepatitis A virus (HAV), or hepatitis C virus (HCV) infection and/or a history of delta virus hepatitis
* Known hypersensitivity or contraindication to any medication or history of allergic reaction to an oligonucleotide or N-acetylgalactosamine (GalNAc)

Additional exclusion criteria for healthy volunteers:

* Evidence of liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-24; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects experiencing adverse events | Part A (SAD phase): through Day 29; Part B (SAD phase): through Day 85; Part C (MAD phase): through Day 176

SECONDARY OUTCOMES:
Profile of Pharmacokinetics (PK) of ALN-HBV | Part A (SAD phase): Day 1; Part B (SAD phase): Day 1; Part C (MAD phase): Days 1 and 85
  Maximum plasma concentration (Cmax)
Profile of Pharmacokinetics (PK) of ALN-HBV | Part A (SAD phase): Day 1; Part B (SAD phase): Day 1; Part C (MAD phase): Days 1 and 85
  Elimination half-life (t1/2)
Profile of Pharmacokinetics (PK) of ALN-HBV | Part A (SAD phase): Day 1; Part B (SAD phase): Day 1; Part C (MAD phase): Days 1 and 85
  Area under the concentration-time curve (AUC)
Change from baseline in quantitative hepatitis B surface antigen (HBsAg) levels | Part B (SAD phase): baseline through Day 85; Part C (MAD phase): baseline through Day 176
  Change in HBsAg levels from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huang, MD, Study Director — Alnylam Pharmaceuticals
Locations (8):
- Australia (3):
  - Clinical Trial Site, Adelaide, South Australia
  - Clinical Trial Site, Fitzroy, Victoria
  - Clinical Trial Site, Parkville, Victoria
- Clinical Trial Site, Hong Kong, Hong Kong
- Clinical Trial Site, Auckland, New Zealand
- Clinical Trial Site, Singapore, Singapore
- Clinical Trial Site, Seoul, South Korea
- Clinical Trial Site, London, United Kingdom

REFERENCES:
- [Derived] Gane E, Lim YS, Kim JB, Jadhav V, Shen L, Bakardjiev AI, Huang SA, Cathcart AL, Lempp FA, Janas MM, Cloutier DJ, Kaittanis C, Sepp-Lorenzino L, Hinkle G, Taubel J, Haslett P, Milstein S, Anglero-Rodriguez YI, Hebner CM, Pang PS, Yuen MF. Evaluation of RNAi therapeutics VIR-2218 and ALN-HBV for chronic hepatitis B: Results from randomized clinical trials. J Hepatol. 2023 Oct;79(4):924-932. doi: 10.1016/j.jhep.2023.05.023. Epub 2023 Jun 7. PMID 37290591